CLINICAL TRIAL: NCT01362595
Title: The Use of Novel Therapies to Reconstitute Blood Cell Production and Promote Organ Performance Using Bone Marrow Failure as a Model: a Pilot, Phase I/II Study of the Amino Acid Leucine in the Treatment of Patients With Transfusion-Dependent Diamond Blackfan Anemia
Brief Title: Pilot Phase I/II Study of Amino Acid Leucine in Treatment of Patients With Transfusion-Dependent Diamond Blackfan Anemia
Acronym: LeucineDBA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Adrianna Vlachos, MD, MD, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-375B
Record Dates: First submitted 2011-05-20; First posted 2011-05-30 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Diamond Blackfan Anemia; Blackfan Diamond Syndrome; DBA; Congenital Hypoplastic Anemia; Pure Red Cell Aplasia
Keywords: leucine administration; red blood cell transfusion; Diamond Blackfan anemia
MeSH Terms: conditions — Anemia, Diamond-Blackfan; Anemia, Hypoplastic, Congenital; Red-Cell Aplasia, Pure | interventions — Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Leucine (Other): No alternative treatment arm
  Interventions: Drug: leucine

INTERVENTIONS:
Drug: leucine — Dosage of leucine will be dependent on body surface area (BSA):
  leucine 700 mg/m2/dose by mouth three times a day
  Other Names: L-leucine

SUMMARY:
This study will determine the safety and possibility of giving the amino acid, leucine, in patients with Diamond Blackfan anemia(DBA)who are on dependent on red blood cell transfusions.

The leucine is expected to produce a response in patients with DBA to the point where red blood cell production is increased. Red cell transfusions can then be less frequent or possibly discontinued.

The investigators will study the side effects, if any, of giving leucine to DBA patients. Leucine levels of leucine will be obtained at baseline and during the study.

The drug leucine will be provided in capsule form and taken 3 times a day for a total of 9 months.

DETAILED DESCRIPTION:
Leucine will be provided to participants in the form of a capsule and will be taken three times daily.

Blood hemoglobin levels will be monitored every 3-4 weeks for 9 months.

The entire study will last 12-15 months in length.

Subjects must be two years of age or older and on transfusion for more than six months prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Diamond Blackfan anemia as published in British Journal of Hematology
* transfusion dependent
* age 2 years and older
* adequate renal function
* adequate liver function
* negative B-HCG if patient is a menstruating female and documentation of adequate contraception
* signed informed consent

Exclusion Criteria:

* Known hypersensitivity to branched chain amino acids
* Diagnosis of an inborn error of amino acid metabolism disorder
* Prior hematopoietic stem cell transplantation
* Pregnancy, or plans to become pregnant during duration of trial

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrianna Vlachos, MD, Principal Investigator — Feinstein Institutes for Medical Research; Cohen Children's Medical Center
Locations (11):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford University Medical Center, Palo Alto, California
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Missouri-Columbia Women's and Children's Hospital, Columbia, Missouri
  - Children's Specialty Center of Nevada, Las Vegas, Nevada
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Draptchinskaia N, Gustavsson P, Andersson B, Pettersson M, Willig TN, Dianzani I, Ball S, Tchernia G, Klar J, Matsson H, Tentler D, Mohandas N, Carlsson B, Dahl N. The gene encoding ribosomal protein S19 is mutated in Diamond-Blackfan anaemia. Nat Genet. 1999 Feb;21(2):169-75. doi: 10.1038/5951. PMID 9988267
- [Background] Gazda HT, Grabowska A, Merida-Long LB, Latawiec E, Schneider HE, Lipton JM, Vlachos A, Atsidaftos E, Ball SE, Orfali KA, Niewiadomska E, Da Costa L, Tchernia G, Niemeyer C, Meerpohl JJ, Stahl J, Schratt G, Glader B, Backer K, Wong C, Nathan DG, Beggs AH, Sieff CA. Ribosomal protein S24 gene is mutated in Diamond-Blackfan anemia. Am J Hum Genet. 2006 Dec;79(6):1110-8. doi: 10.1086/510020. Epub 2006 Nov 2. PMID 17186470
- [Background] Cmejla R, Cmejlova J, Handrkova H, Petrak J, Pospisilova D. Ribosomal protein S17 gene (RPS17) is mutated in Diamond-Blackfan anemia. Hum Mutat. 2007 Dec;28(12):1178-82. doi: 10.1002/humu.20608. PMID 17647292
- [Background] Farrar JE, Nater M, Caywood E, McDevitt MA, Kowalski J, Takemoto CM, Talbot CC Jr, Meltzer P, Esposito D, Beggs AH, Schneider HE, Grabowska A, Ball SE, Niewiadomska E, Sieff CA, Vlachos A, Atsidaftos E, Ellis SR, Lipton JM, Gazda HT, Arceci RJ. Abnormalities of the large ribosomal subunit protein, Rpl35a, in Diamond-Blackfan anemia. Blood. 2008 Sep 1;112(5):1582-92. doi: 10.1182/blood-2008-02-140012. Epub 2008 Jun 5. PMID 18535205
- [Background] Gazda HT, Sheen MR, Vlachos A, Choesmel V, O'Donohue MF, Schneider H, Darras N, Hasman C, Sieff CA, Newburger PE, Ball SE, Niewiadomska E, Matysiak M, Zaucha JM, Glader B, Niemeyer C, Meerpohl JJ, Atsidaftos E, Lipton JM, Gleizes PE, Beggs AH. Ribosomal protein L5 and L11 mutations are associated with cleft palate and abnormal thumbs in Diamond-Blackfan anemia patients. Am J Hum Genet. 2008 Dec;83(6):769-80. doi: 10.1016/j.ajhg.2008.11.004. PMID 19061985
- [Background] Vlachos A, Klein GW, Lipton JM. The Diamond Blackfan Anemia Registry: tool for investigating the epidemiology and biology of Diamond-Blackfan anemia. J Pediatr Hematol Oncol. 2001 Aug-Sep;23(6):377-82. doi: 10.1097/00043426-200108000-00015. PMID 11563775
- [Background] Vlachos A, Federman N, Reyes-Haley C, Abramson J, Lipton JM. Hematopoietic stem cell transplantation for Diamond Blackfan anemia: a report from the Diamond Blackfan Anemia Registry. Bone Marrow Transplant. 2001 Feb;27(4):381-6. doi: 10.1038/sj.bmt.1702784. PMID 11313667
- [Background] Lipton JM, Atsidaftos E, Zyskind I, Vlachos A. Improving clinical care and elucidating the pathophysiology of Diamond Blackfan anemia: an update from the Diamond Blackfan Anemia Registry. Pediatr Blood Cancer. 2006 May 1;46(5):558-64. doi: 10.1002/pbc.20642. PMID 16317735
- [Background] Ozsoylu S. Oral megadose methylprednisolone for Diamond-Blackfan anemia. Blood. 1994 Nov 1;84(9):3245-7. No abstract available. PMID 7949199
- [Background] Bernini JC, Carrillo JM, Buchanan GR. High-dose intravenous methylprednisolone therapy for patients with Diamond-Blackfan anemia refractory to conventional doses of prednisone. J Pediatr. 1995 Oct;127(4):654-9. doi: 10.1016/s0022-3476(95)70134-6. PMID 7562296
- [Background] Buchanan GR; International Diamond-Blackfan Anemia Study Group. Oral megadose methylprednisolone therapy for refractory Diamond-Blackfan anemia. International Diamond-Blackfan Anemia Study Group. J Pediatr Hematol Oncol. 2001 Aug-Sep;23(6):353-6. doi: 10.1097/00043426-200108000-00006. PMID 11563769
- [Background] Totterman TH, Nisell J, Killander A, Gahrton G, Lonnqvist B. Successful treatment of pure red-cell aplasia with cyclosporin. Lancet. 1984 Sep 22;2(8404):693. doi: 10.1016/s0140-6736(84)91245-5. No abstract available. PMID 6147711
- [Background] Williams DL, Mageed AS, Findley H, Ragab AH. Cyclosporine in the treatment of red cell aplasia. Am J Pediatr Hematol Oncol. 1987 Winter;9(4):314-6. doi: 10.1097/00043426-198724000-00007. PMID 3125756
- [Background] Seip M, Zanussi GF. Cyclosporine in steroid-resistant Diamond-Blackfan anaemia. Acta Paediatr Scand. 1988 May;77(3):464-6. doi: 10.1111/j.1651-2227.1988.tb10682.x. PMID 3389144
- [Background] Leonard EM, Raefsky E, Griffith P, Kimball J, Nienhuis AW, Young NS. Cyclosporine therapy of aplastic anaemia, congenital and acquired red cell aplasia. Br J Haematol. 1989 Jun;72(2):278-84. doi: 10.1111/j.1365-2141.1989.tb07695.x. PMID 2503027
- [Background] Splain J, Berman BW. Cyclosporin A treatment for Diamond-Blackfan anemia. Am J Hematol. 1992 Mar;39(3):208-11. doi: 10.1002/ajh.2830390310. PMID 1546717
- [Background] Monteserin MC, Garcia Vela JA, Ona F, Lastra AM. Cyclosporin A for Diamond-Blackfan anemia: a new case. Am J Hematol. 1993 Apr;42(4):406-7. doi: 10.1002/ajh.2830420419. No abstract available. PMID 8493997
- [Background] Alessandri AJ, Rogers PC, Wadsworth LD, Davis JH. Diamond-blackfan anemia and cyclosporine therapy revisited. J Pediatr Hematol Oncol. 2000 Mar-Apr;22(2):176-9. doi: 10.1097/00043426-200003000-00020. PMID 10779036
- [Background] Bobey NA, Carcao M, Dror Y, Freedman MH, Dahl N, Woodman RC. Sustained cyclosporine-induced erythropoietic response in identical male twins with diamond-blackfan anemia. J Pediatr Hematol Oncol. 2003 Nov;25(11):914-8. doi: 10.1097/00043426-200311000-00018. PMID 14608205
- [Background] Harris SI, Weinberg JB. Treatment of red cell aplasia with antithymocyte globulin: repeated inductions of complete remissions in two patients. Am J Hematol. 1985 Oct;20(2):183-6. doi: 10.1002/ajh.2830200212. PMID 3929597
- [Background] Roychowdhury DF, Linker CA. Pure red cell aplasia complicating an ABO-compatible allogeneic bone marrow transplantation, treated successfully with antithymocyte globulin. Bone Marrow Transplant. 1995 Sep;16(3):471-2. PMID 8535322
- [Background] Abkowitz JL, Powell JS, Nakamura JM, Kadin ME, Adamson JW. Pure red cell aplasia: response to therapy with anti-thymocyte globulin. Am J Hematol. 1986 Dec;23(4):363-71. doi: 10.1002/ajh.2830230408. PMID 3098093
- [Background] McGuire WA, Yang HH, Bruno E, Brandt J, Briddell R, Coates TD, Hoffman R. Treatment of antibody-mediated pure red-cell aplasia with high-dose intravenous gamma globulin. N Engl J Med. 1987 Oct 15;317(16):1004-8. doi: 10.1056/NEJM198710153171606. No abstract available. PMID 3116428
- [Background] Bejaoui M, Fitouri Z, Sfar MT, Lakhoua R. Failure of immunosuppressive therapy and high-dose intravenous immunoglobulins in four transfusion-dependent, steroid-unresponsive Blackfan-Diamond anemia patients. Haematologica. 1993 Jan-Feb;78(1):38-9. PMID 8491420
- [Background] Sumimoto S, Kawai M, Kasajima Y, Hamamoto T. Intravenous gamma-globulin therapy in Diamond-Blackfan anemia. Acta Paediatr Jpn. 1992 Apr;34(2):179-80. doi: 10.1111/j.1442-200x.1992.tb00947.x. PMID 1621524
- [Background] Miceli Sopo S, Pesaresi MA, Pastore M, Stabile A. Intravenous immunoglobulin in Diamond-Blackfan anaemia. Eur J Pediatr. 1990 Aug;149(11):779-80. doi: 10.1007/BF01957279. PMID 2226550
- [Background] Halperin DS, Estrov Z, Freedman MH. Diamond-Blackfan anemia: promotion of marrow erythropoiesis in vitro by recombinant interleukin-3. Blood. 1989 Apr;73(5):1168-74. PMID 2649168
- [Background] Dunbar CE, Smith DA, Kimball J, Garrison L, Nienhuis AW, Young NS. Treatment of Diamond-Blackfan anaemia with haematopoietic growth factors, granulocyte-macrophage colony stimulating factor and interleukin 3: sustained remissions following IL-3. Br J Haematol. 1991 Oct;79(2):316-21. doi: 10.1111/j.1365-2141.1991.tb04540.x. PMID 1958491
- [Background] Gillio AP, Faulkner LB, Alter BP, Reilly L, Klafter R, Heller G, Young DC, Lipton JM, Moore MA, O'Reilly RJ. Treatment of Diamond-Blackfan anemia with recombinant human interleukin-3. Blood. 1993 Aug 1;82(3):744-51. PMID 8338944
- [Background] Gillio AP, Faulkner LB, Alter BP, Reilly L, Klafter R, Heller G, Young DC, Lipton JM, Moore MA, O'Reilly RJ. Successful treatment of Diamond-Blackfan anemia with interleukin 3. Stem Cells. 1993 Jul;11 Suppl 2:123-30. doi: 10.1002/stem.5530110820. PMID 7691318
- [Background] Bastion Y, Bordigoni P, Debre M, Girault D, Leblanc T, Tchernia G, Ball S, McGuckin C, Gordon-Smith EC, Bekassy A, et al. Sustained response after recombinant interleukin-3 in diamond blackfan anemia. Blood. 1994 Jan 15;83(2):617-8. No abstract available. PMID 8286756
- [Background] Olivieri NF, Feig SA, Valentino L, Berriman AM, Shore R, Freedman MH. Failure of recombinant human interleukin-3 therapy to induce erythropoiesis in patients with refractory Diamond-Blackfan anemia. Blood. 1994 May 1;83(9):2444-50. PMID 8167334
- [Background] Ball SE, Tchernia G, Wranne L, Bastion Y, Bekassy NA, Bordigoni P, Debre M, Elinder G, Kamps WA, Lanning M, et al. Is there a role for interleukin-3 in Diamond-Blackfan anaemia? Results of a European multicentre study. Br J Haematol. 1995 Oct;91(2):313-8. doi: 10.1111/j.1365-2141.1995.tb05295.x. PMID 8547067
- [Background] Abkowitz JL, Schaison G, Boulad F, Brown DL, Buchanan GR, Johnson CA, Murray JC, Sabo KM. Response of Diamond-Blackfan anemia to metoclopramide: evidence for a role for prolactin in erythropoiesis. Blood. 2002 Oct 15;100(8):2687-91. doi: 10.1182/blood.V100.8.2687. PMID 12351372
- [Background] Akiyama M, Yanagisawa T, Yuza Y, Yokoi K, Ariga M, Fujisawa K, Hoshi Y, Eto Y. Successful treatment of Diamond-Blackfan anemia with metoclopramide. Am J Hematol. 2005 Apr;78(4):295-8. doi: 10.1002/ajh.20278. PMID 15795909
- [Background] Leblanc TM, Da Costa L, Marie I, Demolis P, Tchernia G. Metoclopramide treatment in DBA patients: no complete response in a French prospective study. Blood. 2007 Mar 1;109(5):2266-7. doi: 10.1182/blood-2006-08-039545. No abstract available. PMID 17312003
- [Background] Cynober L, Harris RA. Symposium on branched-chain amino acids: conference summary. J Nutr. 2006 Jan;136(1 Suppl):333S-6S. doi: 10.1093/jn/136.1.333S. No abstract available. PMID 16365109
- [Background] Choudry HA, Pan M, Karinch AM, Souba WW. Branched-chain amino acid-enriched nutritional support in surgical and cancer patients. J Nutr. 2006 Jan;136(1 Suppl):314S-8S. doi: 10.1093/jn/136.1.314S. PMID 16365105
- [Background] Pospisilova D, Cmejlova J, Hak J, Adam T, Cmejla R. Successful treatment of a Diamond-Blackfan anemia patient with amino acid leucine. Haematologica. 2007 May;92(5):e66-7. doi: 10.3324/haematol.11498. No abstract available. PMID 17562599
- [Background] Kimball SR, Jefferson LS. Signaling pathways and molecular mechanisms through which branched-chain amino acids mediate translational control of protein synthesis. J Nutr. 2006 Jan;136(1 Suppl):227S-31S. doi: 10.1093/jn/136.1.227S. PMID 16365087
- [Background] Pencharz PB, Ball RO. Amino acid needs for early growth and development. J Nutr. 2004 Jun;134(6 Suppl):1566S-1568S. doi: 10.1093/jn/134.6.1566S. PMID 15173431
- [Background] Bernardini P, Fischer JE. Amino acid imbalance and hepatic encephalopathy. Annu Rev Nutr. 1982;2:419-54. doi: 10.1146/annurev.nu.02.070182.002223. No abstract available. PMID 6138050
- [Background] Poon RT, Yu WC, Fan ST, Wong J. Long-term oral branched chain amino acids in patients undergoing chemoembolization for hepatocellular carcinoma: a randomized trial. Aliment Pharmacol Ther. 2004 Apr 1;19(7):779-88. doi: 10.1111/j.1365-2036.2004.01920.x. PMID 15043519
- [Background] Plaitakis A, Smith J, Mandeli J, Yahr MD. Pilot trial of branched-chain aminoacids in amyotrophic lateral sclerosis. Lancet. 1988 May 7;1(8593):1015-8. doi: 10.1016/s0140-6736(88)91841-7. PMID 2896868
- [Background] Pass KA, Lane PA, Fernhoff PM, Hinton CF, Panny SR, Parks JS, Pelias MZ, Rhead WJ, Ross SI, Wethers DL, Elsas LJ 2nd. US newborn screening system guidelines II: follow-up of children, diagnosis, management, and evaluation. Statement of the Council of Regional Networks for Genetic Services (CORN). J Pediatr. 2000 Oct;137(4 Suppl):S1-46. doi: 10.1067/mpd.2000.109437. No abstract available. PMID 11044838
- [Background] Vlachos A, Ball S, Dahl N, Alter BP, Sheth S, Ramenghi U, Meerpohl J, Karlsson S, Liu JM, Leblanc T, Paley C, Kang EM, Leder EJ, Atsidaftos E, Shimamura A, Bessler M, Glader B, Lipton JM; Participants of Sixth Annual Daniella Maria Arturi International Consensus Conference. Diagnosing and treating Diamond Blackfan anaemia: results of an international clinical consensus conference. Br J Haematol. 2008 Sep;142(6):859-76. doi: 10.1111/j.1365-2141.2008.07269.x. Epub 2008 Jul 30. PMID 18671700
- [Background] Cmejlova J, Dolezalova L, Pospisilova D, Petrtylova K, Petrak J, Cmejla R. Translational efficiency in patients with Diamond-Blackfan anemia. Haematologica. 2006 Nov;91(11):1456-64. PMID 17082006
- [Background] Hutson SM, Sweatt AJ, Lanoue KF. Branched-chain [corrected] amino acid metabolism: implications for establishing safe intakes. J Nutr. 2005 Jun;135(6 Suppl):1557S-64S. doi: 10.1093/jn/135.6.1557S. PMID 15930469
- [Background] Lab Advisor(TM); Leucine Measurements in Micromedex (R) Healthcare Series. 2010Thomson Reuters
- [Background] Jellin JM, Gregory P, Batz F. Pharmacist's letter/ Prescriber's Letter Natural Medicines Comprehensive Database, 3rd ed, Therapeutic Research Faculty, Stockton, CA, 2000.
- [Background] Braverman ER. The Healing Nutrients Within. New Canaan, CT: Keats Publishing, Inc. 1997; 339
- [Background] Gilman AG, Rall JW, Nies AD et al (eds): Goodman and Gilman's The Pharmacological Basis of Therapeutics, 8th ed. Pergamon Press, New York, NY, 1990.
- [Background] AMA Department of Drugs; AMA Drug Evaluations, 6th ed. American Medical Association, Chicago, IL,1986.
- [Background] Tietz NE (Ed); Clinical Guide to Laboratory Tests, 3rd ed W. B. Saunders, Philadelphia, PA, 1995.
- [Background] Henry JB: Clinical Diagnosis and Management by Laboratory Methods, 20th ed. Saunders 2001.
- [Background] Sax HC, Talamini MA, Fischer JE. Clinical use of branched-chain amino acids in liver disease, sepsis, trauma, and burns. Arch Surg. 1986 Mar;121(3):358-66. doi: 10.1001/archsurg.1986.01400030120019. PMID 3080979
- [Derived] Vlachos A, Atsidaftos E, Lababidi ML, Muir E, Rogers ZR, Alhushki W, Bernstein J, Glader B, Gruner B, Hartung H, Knoll C, Loew T, Nalepa G, Narla A, Panigrahi AR, Sieff CA, Walkovich K, Farrar JE, Lipton JM. L-leucine improves anemia and growth in patients with transfusion-dependent Diamond-Blackfan anemia: Results from a multicenter pilot phase I/II study from the Diamond-Blackfan Anemia Registry. Pediatr Blood Cancer. 2020 Dec;67(12):e28748. doi: 10.1002/pbc.28748. Epub 2020 Oct 6. PMID 33025707
- See also: Diamond Blackfan Anemia Registry - a registry for patients with DBA in North America — http://www.dbar.org
- See also: Daniella Maria Arturi Foundation is a family sponsored group which facilitates research for DBA. — http://www.dmaf.org
- See also: The DBA foundation is a family sponsored organization who raise funds for research and provides emotional support to families. — http://www.dbafoundation.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 subjects were screened and of those 12 did not meet eligibility criteria
Period: Overall Study
Arm/Group | Leucine
Started | 55
Completed | 43
Not Completed | 12
Not completed — Screen failure | 10
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Leucine
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 10.4 [2.5 to 46.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Response to Leucine in Transfusion Dependent Patients With Diamond Blackfan Anemia
Description: The primary outcome is the type of response observed at 9 months. Response to treatment can be one of the following:
  1. Complete response (CR): Hb > 9 gm/dL and transfusion-independence as defined in DBA
  2. Partial response (PR): Hb < 9 gm/dL and increased reticulocyte count to greater than baseline.
  3. No response (NR): no change in transfusion requirements and no significant change reticulocyte count from baseline
  4. Progression: worsening of disease as defined by the need for more frequent transfusions
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Leucine
Number analyzed (Participants) | 43
Participants
  Complete Hematologic Response | 2
  Partial hematologic response | 5
  No hematologic response | 36
  Progression | 0
Statistical Analysis 1: Comparison: Leucine; Test type: Other; Due to the small sample size, the statistical approach is primarily descriptive in nature

2. Secondary Outcome: Severe Adverse Events Attributable to Leucine
Description: Adverse events occurring while participants were on Leucine
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Leucine
Number analyzed (Participants) | 43
Participants
  No Adverse events | 41
  Withdrew early | 2

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Leucine
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT01362595/Prot_SAP_000.pdf